CLINICAL TRIAL: NCT04725513
Title: Pilot Investigation to Evaluate Effectiveness of Shockwave Therapy, a Combination of Shockwave Therapy and Photobiomodulation and Physical Therapy in the Management of Non-insertional Achilles Tendinopathy: A Randomized Control Trial With Elective Cross-Over Design
Brief Title: Pilot Investigation to Evaluate Effectiveness of Shockwave Therapy, Photobiomodulation and Physical Therapy in the Management of Non-insertional Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Adam Tenforde, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000025
Record Dates: First submitted 2021-01-14; First posted 2021-01-26 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Low-Level Light Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: The first part of the study is a randomized control trial, the second part is an elective cross over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Physical Therapy Only (Active Comparator)
  Interventions: Other: Physical Therapy
- Shockwave Therapy and Physical Therapy (Experimental)
  Interventions: Device: Shockwave Therapy; Other: Physical Therapy
- Photobiomodulation, Shockwave Therapy and Physical Therapy (Experimental)
  Interventions: Device: Shockwave Therapy; Device: Photobiomodulation Therapy; Other: Physical Therapy

INTERVENTIONS:
Device: Shockwave Therapy — Participants will receive shockwave therapy once a week for three weeks
  Arms: Photobiomodulation, Shockwave Therapy and Physical Therapy; Shockwave Therapy and Physical Therapy
Device: Photobiomodulation Therapy — Participants will receive photobiomodulation therapy twice a week for three weeks
  Arms: Photobiomodulation, Shockwave Therapy and Physical Therapy
Other: Physical Therapy — Participants will enroll in physical therapy and complete an at-home exercise protocol

SUMMARY:
This is a randomized control trial with an elective cross over after three months to evaluate three different treatments in the management of non-insertional Achilles Tendinopathy. The treatment methods include physical therapy, shockwave therapy and photobiomodulation.

DETAILED DESCRIPTION:
This is a randomized control study with an elective cross over. In part 1 of the study participants will be randomized into one of three treatment arms: 1) physical therapy only; 2) physical therapy and shockwave therapy; 3) physical therapy, shockwave therapy and photobiomodulation. At 3 months, patients can choose to switch to a different treatment arm than they were initially randomized.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of mid-portion Achilles tendinopathy (including both unilateral and bilateral)
* Running is the pre-injury primary form of physical activity and pre-injury would complete on average 10 miles per week or more of running
* VISA-A <80 at baseline to be eligible

Exclusion Criteria

* Less than 3 months of symptoms
* Primary insertional Achilles tendinopathy
* Diagnosis of rheumatological disease/connective tissue condition, symptomatic arthritis of foot and ankle, a primary running related injury outside Achilles tendinopathy, other contraindications to PBMT or SWT
* Have received SWT within the past 3 months to their Achilles
* Prior injection within 3 months
* Currently enrolled in PT for more than 4 weeks for their condition
* Women who are pregnant.
* known history of Achilles tendon tear
* currently taking oral steroid or fluoroquinolone class of antibiotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tenforde AS, Pham L, Gaudette LW, Funk MM, Vogel KE, Bruneau MM, Yuan X, Schroeder JD, Isaacson B, Hagar N, Metzger E, Nolan DC, Tam J, Silbernagel KG. Exercise, radial pressure waves, and photobiomodulation for management of non-insertional Achilles tendinopathy in runners: a three-arm non-blinded randomised control trial. BMJ Open Sport Exerc Med. 2025 Oct 5;11(4):e002442. doi: 10.1136/bmjsem-2024-002442. eCollection 2025. PMID 41070206
- [Derived] Tenforde AS, Vogel KEL, Tam J, Silbernagel KG. Research protocol to evaluate the effectiveness of shockwave therapy, photobiomodulation and physical therapy in the management of non-insertional Achilles tendinopathy in runners: a randomised control trial with elective cross-over design. BMJ Open Sport Exerc Med. 2022 Sep 27;8(3):e001397. doi: 10.1136/bmjsem-2022-001397. eCollection 2022. PMID 36187084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Target enrollment was 60 participants randomly assigned equally to three groups. No power calculations were used to determine sample size as no comparable studies were identified to estimate effects of RPW. Eligible participants were runners aged 18-65 with primary running-related injury diagnosed as unilateral or bilateral non-insertional AT and symptoms exceeding 3 months. Each reported running as their primary sport, with weekly volume >16 km.
Pre-assignment Details: After screening and obtaining written informed consent, participants who enrolled were assigned, using block randomisation design, o one of three conditions: EXER; EXER and RPW; or EXER, RPW and PBMT.
  After 3 months, participants could elect to participate for three additional months using a different treatment than initially prescribed (EXER +RPW or EXER + RPW + PBMT) or could continue EXER and complete a 6-month follow-up visit.
Groups:
- Physical Therapy Only: Participants were all prescribed a four-phase progressive Achilles tendon-loading program. Twice weekly calls were completed over 3 weeks to ensure compliance and answer questions. In addition to the Achilles loading program, each participant was instructed to continue exercises prescribed by their physical therapist to address individual impairments contributing to injury.
- Shockwave Therapy and Physical Therapy: Participants in this treatment arm completed the same loading protocol as EXER and also received RPW delivered once per week for 3 weeks with a telephone check-in later in the week.
- Photobiomodulation, Shockwave Therapy and Physical Therapy: Participants allocated to this treatment protocol completed EXER and also received a combination of RPW and PBMT
Period: enrollment to 3 months
Arm/Group | Physical Therapy Only | Shockwave Therapy and Physical Therapy | Photobiomodulation, Shockwave Therapy and Physical Therapy
Started | 16 | 14 | 16
Completed | 15 | 12 | 15
Not Completed | 1 | 2 | 1
Period: elective cross-over 3 months to 6 months
Arm/Group | Physical Therapy Only | Shockwave Therapy and Physical Therapy | Photobiomodulation, Shockwave Therapy and Physical Therapy
Started | 8 | 14 | 11
Completed | 8 | 14 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Therapy Only | Shockwave Therapy and Physical Therapy | Photobiomodulation, Shockwave Therapy and Physical Therapy | Total
Number analyzed (Participants) | 15 | 12 | 15 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] — age at enrollment
  years | 37 (10) | 42 (13) | 42 (14) | 40 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 7 | 23
  Male | 5 | 6 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 12 | 14 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Calf Raises Performed to Fatigue and Inability to Continue
Description: Calf raises performed to fatigue and inability to continue
Time Frame: Difference from 0-3 months
Measure: Mean (Standard Deviation); unit: Calf raises
Groups:
- Physical Therapy Only: exercise program
- Shockwave Therapy and Physical Therapy: exercise program with three sessions of radial pressure waves
- Photobiomodulation, Shockwave Therapy and Physical Therapy: combination of exercise program, three sessions of radial pressure waves, and 6 sessions of photobiomodulation treatment
Arm/Group | Physical Therapy Only | Shockwave Therapy and Physical Therapy | Photobiomodulation, Shockwave Therapy and Physical Therapy
Number analyzed (Participants) | 15 | 12 | 15
Calf raises | 3 (6) | 8 (13) | 5 (11)

2. Primary Outcome: Ultrasound Measurements in Change of Cross Sectional Area
Description: Changes in the cross-sectional area measured on ultrasound
Time Frame: Difference from 0-3 months
Measure: Mean (Standard Deviation); unit: cross sectional area of tendon in mm^2
Groups:
- Physical Therapy Only: standard exercise program
- Shockwave Therapy and Physical Therapy: exercise program combined with three weekly sessions of radial pressure wave
- Photobiomodulation, Shockwave Therapy and Physical Therapy: exercise program, radial pressure wave for 3 sessions and 6 total PBMT treatments
Arm/Group | Physical Therapy Only | Shockwave Therapy and Physical Therapy | Photobiomodulation, Shockwave Therapy and Physical Therapy
Number analyzed (Participants) | 15 | 12 | 15
cross sectional area of tendon in mm^2 | -0.03 (0.14) | -0.05 (0.06) | -0.03 (0.15)

3. Primary Outcome: Victorian Institute of Sports Assessment (VISA-A) Questionnaire
Description: Victorian Institute of Sports Assessment Questionnaire. The score of the questionnaire ranges from 0-100, where 100 is a person who is completely asymptomatic (better).
Time Frame: change from baseline to 3 month follow-up measure
Measure: Mean (Standard Deviation); unit: VISA-A units on a scale
Arm/Group | Physical Therapy Only | Shockwave Therapy and Physical Therapy | Photobiomodulation, Shockwave Therapy and Physical Therapy
Number analyzed (Participants) | 15 | 12 | 15
VISA-A units on a scale | 18 (17) | 33 (15) | 25 (40)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Both expected and unexpected changes in health were recorded as adverse events and were obtain after each treatment and at each follow-up timepoint
Arm/Group | Physical Therapy Only | Shockwave Therapy and Physical Therapy | Photobiomodulation, Shockwave Therapy and Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 10/16 | 10/14 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Therapy Only (N=16) | Shockwave Therapy and Physical Therapy (N=14) | Photobiomodulation, Shockwave Therapy and Physical Therapy (N=16)
Expected adverse event defined as pain, soreness, bruising or swelling (Musculoskeletal and connective tissue disorders) | 10 (13) | 10 (14) | 9 (11) — all were reported as mild to moderate, these were obtained from baseline to 3 months of the initial intervention study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04725513/Prot_SAP_003.pdf
  • Informed Consent Form (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT04725513/ICF_000.pdf